CLINICAL TRIAL: NCT05024097
Title: A Phase I-II Study to Test the Safety and Efficacy of PD1 (AB122) and Adenosine Receptor (AB928) Antagonists With Chemotherapy After Short-Course Radiation for Rectal Cancer.
Acronym: PANTHER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-02023289
Record Dates: First submitted 2021-08-20; First posted 2021-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Folfox protocol; zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation therapy and etrumadenant (AB928) (Experimental): Enrolled patients will receive Radiation therapy of 25 Gy in 5 fractions along with etrumadenant 150mg oral drug taken once daily. this will then be followed by 9 cycles of FOLFOX in combination of etrumadenant and zimberelimab investigational drugs.
  Interventions: Drug: Etrumadenant (AB928); Radiation: Radiation therapy; Drug: FOLFOX regimen; Drug: Zimberelimab (AB122)

INTERVENTIONS:
Drug: Etrumadenant (AB928) — Patients will receive a radiation therapy dose of 25Gy in 5 fractions in combination with etrumadenant 150 mg orally, once daily as part of a continuous dose regimen.
Radiation: Radiation therapy — Patients will receive a radiation therapy dose of 25Gy in 5fx
Drug: FOLFOX regimen — After completing the radiation therapy, patients will receive FOLFOX regimen for 9 cycles in combination with etrumadenant and zimberelimab. All patients will be offered adjuvant zimberelimab for up to one year.
Drug: Zimberelimab (AB122) — After completing the radiation therapy, patients will receive FOLFOX regimen for 9 cycles in combination with etrumadenant and zimberelimab. All patients will be offered adjuvant zimberelimab for up to one year.

SUMMARY:
Enrolled patients will receive upfront (week 1) short-course radiotherapy to gross pelvic disease (25Gy in 5fx) in combination with AB928 (150 mg orally, once daily as part of a continuous dose regimen). This will be followed by consolidation chemotherapy (weeks 3-20) with mFOLFOX x9 cycles in combination with AB928 and AB122.

DETAILED DESCRIPTION:
Enrolled patients will receive upfront (week 1) short-course radiotherapy to gross pelvic disease (25Gy in 5fx) in combination with AB928 (150 mg orally, once daily as part of a continuous dose regimen). This will be followed by consolidation chemotherapy (weeks 3-20) with mFOLFOX x9 cycles in combination with AB928 and AB122. Patients will thereafter be assessed for therapeutic responses (week 22-24) with a digital rectal examination, pelvic MRI, and endoscopy. Each case will be reviewed by the Weill Cornell Medicine Colorectal Multidisciplinary Tumor Board for consensus agreement regarding clinical treatment response. The patients thereafter will proceed with total mesorectal excision (TME, week 24) by transabdominal resection for pathologic evaluation (primary tumor and pelvic lymph nodes will be examined).

ELIGIBILITY:
Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen should be included.

Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the rectum
* Age ≥ 18 years
* ECOG performance status 0-1
* cT3N0 or cT1-3N1 or cT4 or cN2
* 5cm from the anal verge
* Rectal cancer amenable to total mesorectal excision
* No evidence of distant metastases
* No prior pelvic radiation therapy
* No prior chemotherapy or surgery for rectal cancer
* No infections requiring systemic antibiotic treatment
* Hgb >8.0 gm/dL, PLT > 150,000/mm3, total bilirubin ≤ 1.5x upper limit of normal, AST ≤ upper limit of normal, ALT ≤ 3x upper limit of normal
* Patients must read, agree to, and sign a statement of informed consent prior to participation in this study. Patients who do not read or understand English or eligible but must have the consent form bread to them in its entirety by an official translator. Informed consent for non-literate or non-English speaking patients may not be obtained by using a relative or a member of the patient's clinical team as a translator
* Female participants or reproductive potential, defined as not surgically sterilized and between menarche and 1 year post menopause, must have a negative serum pregnancy test within 4 weeks prior to initiation of study treatment
* Female participants of reproductive potential and male participants with female partners of reproductive potential must remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive measures from the start of study treatment until 30 days after the last dose of Etrumadenant, -120 days after the last dose of Zimberelimab, whichever is longer and duration of contraception to follow oxaliplatin should be at least 9 months after the last dose for women and 6 months after the last dose for men)
* Women with childbearing potential who are negative for pregnancy (urine or blood) and who agree to use effective contraceptive methods. A woman of childbearing potential is defined by one who is biologically capable of becoming pregnant. Reliable contraception should be used from trial screening and must be continued throughout the study.
* Male subjects must also agree to use effective contraception.

Exclusion Criteria:

* Recurrent rectal cancer
* Primary unresectable rectal cancer is defined as a primary rectal tumor which, on the basis of either physical exam or pelvic MRI, is demed to be adherent or fixed to adjacent pelvic structures (en bloc resection wll not be achieved with negative margins).
* Involved radial margin
* Serum creatinine level >1.5x the upper limit of normal
* Patients who have received prior pelvic radiotherapy
* QTc ≥480 msec using Fredericia's QT correction formula
* Due to the potential risk for drug-drug interactions with etrumadenant, participants must not have had:

  * Treatment with known BCRP substrates with a narrow therapeutic window, administered orally (e.g., prazosin, rosuvastatin) within 4 weeks or 5 half-lives of the drug (whichever is shorter) prior to initiation of and throughout study treatment
  * Treatment with known P-gp substrates with a narrow therapeutic window, administered orally (e.g., digoxin) within 4 weeks or 5 half-lives of the drug (whichever is shorter) prior to initiation of study treatment
  * Treatment with known strong CYP3A4 inducers (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort) and strong CYP3A4 inhibitors (e.g., clarithromycin, grapefruit juice, itraconazole, ketoconazole, posaconazole, telithromycin, and voriconazole) within 4 weeks (for investigational drugs when half- life is unknown or not accurately determined) or 5 drug-elimination half-lives of the drug (when half-life is determined), whichever is longer, or if it is a marketed drug, then 5 drug-elimination half-lives of the drug, prior to initiation of study treatment
  * Refer to the following for more examples of relevant substrates, inhibitors, and inducers with the potential for drug-drug interactions with Etrumadenant: https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug- interactions-table-substrates-inhibitors-and- Inducers
  * Patients receiving herbal and natural remedies. Concomitant use of therapies that contain cannabinoids may be permitted based on the Investigator's discretion.
  * Sensitive substrates of BSEP, MATE1and OCT2.
* Any gastrointestinal condition that would preclude the use of oral medications (e.g., difficulty swallowing, nausea, vomiting, or malabsorption)
* Prior treatment with an agent targeting the adenosine pathway
* Patients with prior allogenic stem cell or solid organ transplantation
* Any active autoimmune disease or a documented history of autoimmune disease or syndrome that required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs), except for vitiligo or resolved childhood asthma/atopy
* Patients with history of idiopathic pulmonary fibrosis, pneumonitis, or interstitial lung disease
* Patients receiving treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor-α agents) administered at >10 mg/day prednisone or equivalent within 2 weeks prior to initiation of study treatment
* Patients who received a live vaccine within 30 days
* Patients who are known to have dihydropyrimidine dehydrogenase (DPD) deficiency
* Patients with peripheral neuropathy Grade ≥ 2
* History of severe allergic reactions to chimeric or humanized antibodies or fusion proteins
* Patients with a history of any arterial thrombitic event within the past 6 months,
* Patients with any other concurrent medical or psychiatric condition or disease which, in the investigator's judgment would make them inappropriate candidates for entry into this study
* Patients with a history of prior malignancy within the past 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer.
* Patients with a history of thrombotic episodes, such as deep venous thrombosis, pulmonary embolus, MI or CVA occurring more than 6 months prior to enrollment may be considered for protocol participation, provided they are on stable doses of anticoagulant therapy. Patients who are anticoagulated for atrial fibrillation or other conditions may participate, provided they are on stable doses of anticoagulant therapy.
* Patients receiving other anticancer or experimental therapy. No other experimental therapies (including chemotherapy, radiation, hormonal treatment, antibodiy therapy, immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, matrix metalloprotease inhibitors, thalidomide, anti-VEGF/Flk-1 monoclonal antibody, or other experimental drugs) of any kind are permitted while the patient is receiving study treatment.
* Women who are pregnant or breastfeeding. Women of childbearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for up to four weeks after the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of treated patients who achieve complete pathologic response | Week 24
  The primary endpoint is the proportion of treated rectal cancer patients who achieve a complete pathologic response.
  All patients will be offered surgical resection however those who achieve a clinical CR at the time of clinical response assessment may choose a non-operative management approach. Due to practicality the latter will be included as complete responders at the time of analysis for this trial.

SECONDARY OUTCOMES:
Number of patients who experience treatment-related adverse events | Day 5 of radiation therapy
  Number of patients with treatment-related early and late adverse events as assessed by the CTCAE version 5.0
Number of patients who experience treatment-related adverse events | 3 months
  Number of patients with treatment-related early and late adverse events as assessed by the CTCAE version 5.0
Number of patients who experience treatment-related adverse events | 6 months
  Number of patients with treatment-related early and late adverse events as assessed by the CTCAE version 5.0
Number of patients who experience treatment-related adverse events | 12 months
  Number of patients with treatment-related early and late adverse events as assessed by the CTCAE version 5.0
Number of patients who experience treatment-related adverse events | 60 months
  Number of patients with treatment-related early and late adverse events as assessed by the CTCAE version 5.0
Progression free survival | 36 months
  PFS is defined as the duration of time from start of treatment to time of progression.
Overall survival | 60 months
  Overall Survival is defined as the duration of time from start of treatment until death.

CONTACTS AND LOCATIONS:
Overall Officials: Encouse Golden, M.D., Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Weill Cornell Medical College, New York, New York
  - Brooklyn Methodist Hospital - NewYork Presbyterian, New York, New York
  - New York Presbyterian Hospital - Queens, New York, New York

IPD SHARING:
Plan to Share IPD: No